CLINICAL TRIAL: NCT05265000
Title: Transcutaneous Spinal Cord Stimulation for Chronic Low Back Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Science Foundation Center for Disruptive Musculoskeletal Innovations (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: tSCS4LBP
Record Dates: First submitted 2022-02-22; First posted 2022-03-03 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Chronic Low-back Pain
Keywords: non-invasive, spinal cord stimulation, neuromodulation

STUDY DESIGN:
Masking Description: Individuals performing the analysis will be blinded to the condition (baseline vs. post therapy)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- tSpinalStim (Experimental): Individuals in this arm will receive spinal cord stimulation
  Interventions: Device: tSpinalStim

INTERVENTIONS:
Device: tSpinalStim — Patients will undergo 12-21 sessions of spinal cord stimulation therapy (30 minutes per session, 3 times a week). Up to five round stimulating electrodes will be placed on the skin midline between spinous processes in cervical, thoracic and/or lumbar region, as cathodes and rectangular pads will be placed symmetrically on the skin over the iliac crests as anodes. The stimulator generates pain-free biphasic rectangular waveform with 1 ms width pulses filled with 5-10 kHz (kilohertz) carrier frequency. A range of stimulation intensities from 0-250 mA (milliamps) may be used. We expect that the stimulation intensities needed for therapeutic effect may differ based on individual's body mass index and/or the amount of subcutaneous fat present at the stimulation site.
  Other Names: Transcutaneous spinal cord stimulation

SUMMARY:
As a leading cause of disability worldwide, chronic low back pain (cLBP) represents a significant medical and socioeconomic problem with estimated health care spending of $87 billion/annually. The efficacy of dorsal column electrical stimulation to inhibit pain was first described over 50 years ago. Since then, several large clinical trials have investigated the therapeutic potential of electrical spinal cord stimulation (SCS) and found that over 70% of patients with intractable pain had over 50% pain relief after 1 year of treatment. Thus, SCS is a promising therapeutic intervention that has superior patient outcomes when compared to traditional modalities for the treatment of cLBP. To date, SCS for treatment of cLBP has been delivered via epidural electrodes, requiring neurosurgical implantation. Although, the implantable stimulators have a low rate of adverse events, secondary complications associated with surgical intervention still occur.Transcutaneous spinal cord stimulation (tSCS) is a rapidly developing non invasive neuromodulation technique in the field of spinal cord injury. Its application potentiates lumbosacral spinal cord excitability enabling motor functions, (e.g. independent standing, postural control) in patients with chronic complete motor paralysis. Given that epidural and transcutaneous SCS activate similar neuronal networks, tSCS for cLBP treatment may be advantageous due to its non-invasive nature which may also allow for a mass market production and rapid patient availability if tSCS is proven efficacious. In this pilot study we will establish the feasibility of tSCS to acutely improve patient reported outcomes (pain scores) and several objective measures, including sit-to-stand biomechanics, neurophysiological and neuroimaging outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Low back pain
* Able to get in and out of chair unassisted
* No changes in medication within 2 weeks of study enrollment
* Stable dose of their medications within 2 weeks of study enrollment

Exclusion Criteria:

* Body Mass Index (BMI) > 28
* Hardware in the spine from prior surgeries
* Presence of epidural stimulation leads
* Presence of any additional neuromuscular pain unrelated to spinal condition
* Intolerance to any form of electrical stimulation, such as neuromuscular stimulation in the past
* Lack of perceived endurance to go through multiple experimental assessments in one day/complete the study which may take up to 3 hours
* Changes in medications within 2 weeks of study enrollment
* Moderate/severe depression (Beck Depression Inventory score > 20)

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) score | 3 hours
  A patient reported outcome of pain; will be assessed by presenting a VAS tool with the scale of 0 -10, 0 - being no pain and 10 the worst pain imaginable. VAS scores will be collected before and after the intervention
Max Sagittal Vertical Axis | 3 hours
  A kinematic variable that measures body flexion (degrees) relative to the vertical sagittal axis (virtual straight line through the midline of the body) assessed using Kinect-2 depth camera while subject performs 3-5 trials of sit-to-stand movement
L5S1/Torso Max Flex/Ext angle | 3 hours
  A kinematic variable that measures torso/L5S1 joint flexion and extension (degrees) assessed using Kinect-2 depth camera while subject performs 3-5 trials of sit-to-stand movement. The maximum flexion and extension will be compared between baseline and post-intervention.
L5S1/Torso Max velocity | 3 hours
  A kinetic variable that measures torso/L5S1 velocity (m/s) assessed using Kinect-2 depth camera while subject performs 3-5 trials of sit-to-stand movement. The maximum velocities will be compared between baseline and post-intervention.
Hip/Pelvis Max Flex/Ext angle | 3 hours
  A kinematic variable that measures pelvis/hip joint flexion and extension (degrees) assessed using Kinect-2 depth camera while subject performs 3-5 trials of sit-to-stand movement The maximum flexion and extension will be compared between baseline and post-intervention.
Hip/Pelvis Max velocity | 3 hours
  A kinematic variable that measures pelvis/hip joint velocity (m/s) assessed using Kinect-2 depth camera while subject performs 3-5 trials of sit-to-stand movement The maximum velocity will be compared between baseline and post-intervention.
Thing/Knee Max Flex/Ext angle | 3 hours
  A kinetic variable that measures thigh/knee joint flexion and extension (degrees) assessed using Kinect-2 depth camera while subject performs 3-5 trials of sit-to-stand movement The maximum flexion and extension will be compared between baseline and post-intervention.
Thing/Knee Max Velocity | 3 hours
  A kinetic variable that measures thigh/knee joint velocity (m/s) assessed using Kinect-2 depth camera while subject performs 3-5 trials of sit-to-stand movement The maximum flexion and extension will be compared between baseline and post-intervention.
Insula - Cingulate connectivity | 3 hours
  A neuroimaging outcome variable that measures functional connectivity (Fisher z-scores, Fz) between the Insula - and Cingulate brain regions. Patients will undergo brain functional magnetic resonance imaging (fMRI) scan before and after intervention. Fz scores will be compared between baseline and post-intervention
Default Mode Network connectivity | 3 hours
  A neuroimaging outcome variable that measures functional connectivity (Fisher-z scores, Fz) of the brain default mode network. Patients will undergo brain functional magnetic resonance imaging (fMRI) fMRI scan before and after intervention. Fz scores will be compared between baseline and post-intervention
Erector Spinae activation (Root Mean Square) | 3 hours
  Erector Spinae (ES) activation will be measured using surface electromyography (EMG) recorded with bilateral EMG electrodes placed at L5 levels while patient performs 3-5 trials of sit-to-stand (concomitant with biomechanics assessment). The root mean square will be calculated during the time period it take the patient to completed sit-to-stand transition (from lift off from the chair to standing)
Rectus Femoris activation (Root Mean Square) | 3 hours
  Rectus femoris (ES) activation will be measured using surface electromyography (EMG) recorded with bilateral EMG electrodes placed on top of the muscle belly at mid thigh while patient performs 3-5 trials of sit-to-stand (concomitant with biomechanics assessment). The root mean square will be calculated during the time period it take the patient to completed sit-to-stand transition (from lift off from the chair to standing)

SECONDARY OUTCOMES:
Shank/Ankle Max Flex/Ext angle | 3 hours
  A kinematic variable that measures shank/ankle joint flexion and extension (degrees) assessed using Kinect-2 depth camera while subject performs 3-5 trials of sit-to-stand movement The maximum flexion and extension will be compared between baseline and post-intervention.
Shank/Ankle Max velocity | 3 hours
  A kinetic variable that measures shank/ankle joint velocity (m/s) assessed using Kinect-2 depth camera while subject performs 3-5 trials of sit-to-stand movement The maximum velocity will be compared between baseline and post-intervention.
Erector Spinae activation (Root Mean Square) | 3 hours
  Erector Spinae (ES) activation will be measured using surface electromyography (EMG) recorded with bilateral EMG electrodes placed at T10 levels while patient performs 3-5 trials of sit-to-stand (concomitant with biomechanics assessment). The root mean square will be calculated during the time period it take the patient to completed sit-to-stand transition (from lift off from the chair to standing)

CONTACTS AND LOCATIONS:
Overall Officials: Anastasia Keller, PhD, Principal Investigator — University of California, San Francisco; Jeannie Bailey, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- San Francisco VA Medical Center, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified raw data will be deposited in a publically available data repository and/or can be made available per request to the principal investigators of the study
Supporting Information: Study Protocol, CSR, Analytic Code
Time Frame: The data will be available after all data has been collected and analyzed and will be available indefinitely.
Access Criteria: Anyone may send a request to the principal investigators for the deidentified participant data to be shared with them. Anyone who has access to the internet/data repositories may access the publicly deposited de-identified participant data.

REFERENCES:
- See also: If you are interested in participating in the study, please follow the link to the initial patient screening survey — https://ucsf.co1.qualtrics.com/jfe/form/SV_0oYFlZbwWwOgOOy